CLINICAL TRIAL: NCT06196294
Title: GPC3/Mesothelin Targeted CAR-γδT for Immunotherapy of Solid Cancer: Phase I Clinical Trial
Brief Title: GPC3/Mesothelin-CAR-γδT Cells Against Cancers
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Second Affiliated Hospital of Guangzhou Medical University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZZCAR-γδT-019
Record Dates: First submitted 2023-12-22; First posted 2024-01-09 (Actual); Last update posted 2024-06-26 (Actual); Status verified 2024-06

CONDITIONS: Pancreas Cancer; Lung Cancer; Liver Cancer; Mesothelioma; CAR-T Cell Therapy; Solid Tumor, Adult
Keywords: Solid Tumor; CAR-γδT; γδT; GPC3; Mesothelin
MeSH Terms: conditions — Pancreatic Neoplasms; Lung Neoplasms; Liver Neoplasms; Mesothelioma | interventions — Cell- and Tissue-Based Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- γδT cell therapy for solid tumor (Experimental)
  Interventions: Biological: Cell therapy for solid tumors
- CAR-γδT cell therapy for solid tumor (Experimental)
  Interventions: Biological: Cell therapy for solid tumors

INTERVENTIONS:
Biological: Cell therapy for solid tumors — Transfer γδT cells into patients for anti-ancer therapy.

SUMMARY:
The third generation of GPC3/mesothelin targeted CAR-γδT cells have been constructed and their anti-cancer function has been verified by multiple in vitro and in vivo studies. Clinical studies will be performed to test anti-cancer function of the CAR-γδT cells for immunotherapy of human cancer patients with GPC3 or Mesothelin expressions. In this phase I study, the safety, tolerance, and preliminary efficacy of the GPC3/Mesothelin-CAR-γδT cell immunotherapy on human cancers will firstly be evaluated.

DETAILED DESCRIPTION:
1. Choose appropriate patients with advanced solid cancers, with written consent for this study;
2. Perform biopsy to determine the expression of GPC3 or Mesothelin of the tumors by western blotting or IHC;
3. Collect blood from the patients and isolate mononuclear cells, select and grow γδT cells and transfect the γδT cells with GPC3 or Mesothelin targeting CAR, amplify the transfected γδT cells as needed, test the quality and killing activity of the CAR-γδT cells and then transfer them back the patients via systemic or local injections, and follow up closely to collect related results as required;
4. To enhance the killing capability, cotreatment the patients with PD1/PDL1/CTLA4 antibodies may be applied;
5. Evaluate the clinical results as needed.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with advanced cancer that expresses GPC3 or Mesothelin protein; 2. Life expectancy >12 weeks; 3. Adequate heart, lung, liver, kidney, and blood function; 4. Available autologous transduced T cells with greater than or equal to 20% expression of GPC3/Mesothelin-CAR determined by flow-cytometry and killing of Mesothelin-positive targets greater than or equal to 20% in cytotoxicity assay; 5. Informed consent explained to, understood by and signed by patient/guardian. Patient/guardian given copy of informed consent.

-

Exclusion Criteria:

1. Had accepted gene therapy before;
2. Severe virus infection such as HBV, HCV, HIV, et al;
3. Known HIV positivity;
4. Active infectious disease related to bacteria, virus,fungi,et al;
5. Other severe diseases that the investigators consider not appropriate;
6. Pregnant or lactating women;
7. Systemic steroid treatment (greater than or equal to 0.5 mg prednisone equivalent/kg/day);
8. Other conditions that the investigators consider not appropriate. -

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-05-10 (Actual); Primary Completion 2030-11-30 (Estimated); Study Completion 2036-12-30 (Estimated)

PRIMARY OUTCOMES:
Number of Patients with Dose Limiting Toxicity | Six months
  A dose limiting toxicity is defined as any toxicity that is considered to be primarily related to the γδT cells, which is irreversible, or life threatening or hematologic or non-hematologic Grade 3-5.

SECONDARY OUTCOMES:
Percent of Patients with best response as either complete remission or partial remission. | Six months
  Response rates will be estimated as the percent of patients whose best response is either complete remission or partial remission by combining the data from the patients. To compare with historical data, a 95% confidence interval will be calculated for the response rate.
Median γδT cell persistence | Six years
  Median γδT cell persistence will be measured by quantitative rt-PCR.

CONTACTS AND LOCATIONS:
Overall Officials: Zhenfeng Zhang, MD, PhD, Principal Investigator — Second Affiliated Hospital of Guangzhou Medical University
Locations (1):
- The Second Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No